CLINICAL TRIAL: NCT03795701
Title: To Predict Weight Loss Response to Liraglutide (Saxenda®), From fMRI-based Determination of Food Cue Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Martin Binks, Associate Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTUIRB2018-824
Record Dates: First submitted 2018-12-17; First posted 2019-01-08 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Obesity
Keywords: Neuroimaging; Hormones
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects in placebo group will receive placebo plus behavioral weight loss counselling to portion control to achieve 500 kcal daily deficit based on MedGem required maintenance calories (not to be reduced below 1000 kcal per day for any subject). Subjects will also be asked to maintain physical activity.
  Interventions: Other: Placebo
- Liraglutide 3.0 (Experimental): Subjects in Liraglutide 3.0 group will receive Saxenda® plus behavioral weight loss counselling to portion control to achieve 500 kcal daily deficit based on MedGem required maintenance calories (not to be reduced below 1000 kcal per day for any subject). Subjects will be asked to maintain physical activity. The dose of Saxenda® will be increased weekly in the first 4 weeks (.6; 1.2; 1.8; 2.4 mg) and maintained on 3 mg for 12 weeks.
  Interventions: Drug: Saxenda®

INTERVENTIONS:
Drug: Saxenda® — Receiving escalating dose of Saxenda® for the first 4 weeks (0.6mg, 1.2mg, 1.8mg, 2.4 mg) and receiving full-dose (3.0 mg) for 12 weeks.
  Other Names: Liraglutide 3.0
  Arms: Liraglutide 3.0
Other: Placebo — Receiving equivalent volumes of the pre-filled solutions from pen-injector as Liraglutide 3.0 group .
  Arms: Placebo

SUMMARY:
The study is a single center, randomized, double blind, placebo controlled; parallel-group repeated measures design. Subjects will be randomly assigned to either Saxenda® or placebo group after baseline assessments. The study will consist of a 4-week partial dose period (Liraglutide 0.6mg, 1.2mg, 1.8mg, 2.4 mg) and a 12-week full-dose (Liraglutide 3.0 mg) period. The placebo group will administer equivalent volumes of the pre-filled solutions from pen-injector at the same time, using the same method during this period. The study proposes to identify factors contributing to early weight loss response in a Saxenda® treatment program. Specifically, the proposed experiments will help determine if Saxenda® changes brain functional Magnetic Resonance Imaging Food Cue Reactivity (fMRI-FCR) and whether the magnitude of that change is associated with changes in behavioral and physiological variables (hunger, satiety, cravings and weight loss).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* BMI 30-50 kg/m2

Exclusion Criteria:

* Participants unable or unwilling to provide informed consent.
* Participants with motor, visual or hearing impairment.
* Females with irregular menstrual cycles (onset of menstruation greater than 1 week from expected data during the last 3 months).
* Females who are currently breastfeeding or intend to start breastfeeding.
* Participants with diagnosed diabetes mellitus (type 1 or type 2) or uncontrolled hypertension, history of ischemic heart disease, stroke, neurological disease.
* Participants with current severe psychiatric illnesses (e.g. psychosis, schizophrenia, bipolar disorders, depression).
* Participants experiencing current suicidal ideation, and recent or past suicide attempts.
* Participants with history of psychiatric hospitalization.
* Participants who are currently on (or have been on within the past 4 weeks) any medication in the broader drug classes of anti-depressant, anti-epileptic, or anti-anxiety medicines will be excluded (as these affect fMRI-FCR in the brain).
* Participants with contraindications for MRI scanning.

  1. aneurism clips
  2. any implanted medical devices (pacemaker, neurostimulator)
  3. known pregnancy
  4. shrapnel in body or any injury to eye involving metal
  5. any ferrous metal in body
* Participants with a history of diagnosed eating disorders such as bulimia nervosa, anorexia nervosa and severe binge eating disorder.
* Participants with a history of diagnosed substance abuse or alcohol abuse.
* Patients experiencing persistent loss of appetite, nausea or vomiting within the last 4 weeks without known cause (e.g. flu, food poisoning).
* Participants who have been involved in a weight loss intervention program (including anti-obesity medication) within the past 3 months (and or loss >10% of body weight) or who have ever had bariatric surgery or have weight loss devices implanted.
* Current smokers (smoked within the last 30 days).
* The receipt of any investigational drug within (3 months) prior to this trial.
* Previous participation in this trial (i.e. randomized).
* Unable or unwilling to consume required study meals for any reason (e.g. dietary restrictions, allergies, or aversions to any of the food items used in the study).
* Contraindications to study medications,

  * Subject with a personal or family history of medullary thyroid carcinoma (MTC).
  * Subject with multiple endocrine neoplasia syndrome 2 (MEN 2).
  * Allergic to Liraglutide or any of the ingredients in Saxenda® (i.e. Active ingredient: liraglutide; Inactive ingredients: disodium phosphate dehydrate, propylene glycol, phenol and water for injection)
  * Women who are pregnant, or have the intention of becoming pregnant.
* Taking other GLP-1 receptor agonists (currently or in the past 3 months).
* Current severe problems with stomach, such as slowed emptying of the stomach (gastroparesis) or problems with digesting food.
* Current or past known serious chronic illness of liver, kidney and pancreas.
* Current or recent (30 days) depression or suicidal thoughts.
* Current fasting plasma glucose 126mg/dL or higher or HbA1c 6.5% or higher, or alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine, blood urea nitrogen (BUN) 10% above normal range for the assay.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Compare the changes of pre-prandial fMRI-FCR in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Pre-prandial fMRI-FCR will be measured via fMRI
Compare the changes of post-prandial fMRI-FCR in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Post-prandial fMRI-FCR will be measured via fMRI
Compare the changes of energy intake in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Energy intake will be assessed via ad libitum feeding
Compare the changes of hunger/satiety in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Hunger/satiety will be assessed via Visual Analog Scale (VAS). Subjects will rate on the 100 mm line with a vertical line. There is no specific number on the scale. On each 100-mm line, an sensation is paired with the opposing sensation, (for example, 'not at all hungry' and 'extremely hungry' or 'Not at all satiated' and 'extremely satiated').
Compare the changes of hunger/satiety in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Hunger/satiety will be assessed via glucagon-like peptide-1 (GLP-1)
Compare the changes of hunger/satiety in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Hunger/satiety will be assessed via Peptide YY (PYY)
Compare the changes of hunger/satiety in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Hunger/satiety will be assessed via ghrelin
Prediction of weight loss in Liraglutide 3.0 group by examine early change in pre-prandial fMRI-FCR | Baseline, Week 4, and Week 16
  Pre-prandial fMRI-FCR will be measured via fMRI
Prediction of weight loss in Liraglutide 3.0 group by examine early change in post-prandial fMRI-FCR | Baseline, Week 4, and Week 16
  Post-prandial fMRI-FCR will be measured via fMRI

SECONDARY OUTCOMES:
Correlation between changes in post-prandial fMRI-FCR and changes in energy intake | Baseline, Week 4, and Week 16
  Post-prandial fMRI-FCR measured via fMRI. Energy intake will be assessed via ad libitum feeding.
Correlation between changes in post-prandial fMRI-FCR and changes in hunger/satiety | Baseline, Week 4, and Week 16
  Post-prandial fMRI-FCR measured via fMRI. Hunger/satiety will be measured via Visual Analog Scale (VAS). Subjects will rate on the 100 mm line with a vertical line. There is no specific number on the scale. On each 100-mm line, an sensation was paired with the opposing sensation, (for example, 'not at all hungry' and 'extremely hungry').
Correlation between changes in post-prandial fMRI-FCR and changes in hunger/satiety | Baseline, Week 4, and Week 16
  Post-prandial fMRI-FCR measured via fMRI. Hunger/satiety will be measured via glucagon-like peptide-1 (GLP-1).
Correlation between changes in post-prandial fMRI-FCR and changes in hunger/satiety | Baseline, Week 4, and Week 16
  Post-prandial fMRI-FCR measured via fMRI. Hunger/satiety will be measured via peptide YY (PYY).
Correlation between changes in post-prandial fMRI-FCR and changes in hunger/satiety | Baseline, Week 4, and Week 16
  Post-prandial fMRI-FCR measured via fMRI. Hunger/satiety will be measured via ghrelin.
Examine if the correlations described in outcome 10 differ in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Energy intake will be assessed via ad libitum feeding.
Examine if the correlations described in outcome 11 differ in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Hunger/satiety will be measured via Visual Analog Scale (VAS). Subjects will rate on the 100 mm line with a vertical line. There is no specific number on the scale. On each 100-mm line, an sensation was paired with the opposing sensation, (for example, 'not at all hungry' and 'extremely hungry').
Examine if the correlations described in outcome 12 differ in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Hunger/satiety will be measured via glucagon-like peptide-1 (GLP-1)
Examine if the correlations described in outcome 13 differ in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Hunger/satiety will be measured via peptide YY (PYY)
Examine if the correlations described in outcome 14 differ in Liraglutide 3.0 vs. Placebo Group | Baseline, Week 4, and Week 16
  Hunger/satiety will be measured via ghrelin
Prediction of weight loss after 16 weeks intervention by assessing early changes in energy intake | Baseline, Week 4, and Week 16
  Energy intake will be assessed via ad libitum feeding
Prediction of weight loss after 16 weeks intervention by assessing early changes in hunger/satiety | Baseline, Week 4, and Week 16
  Hunger/satiety will be measured via Visual Analog Scale (VAS). Subjects will rate on the 100 mm line with a vertical line. There is no specific number on the scale. On each 100-mm line, an sensation was paired with the opposing sensation, (for example, 'not at all hungry' and 'extremely hungry' or 'Not at all satiated' and 'extremely satiated').
Prediction of weight loss after 16 weeks intervention by assessing early changes in hunger/satiety | Baseline, Week 4, and Week 16
  Hunger/satiety will be measured via glucagon-like peptide-1 (GLP-1)
Prediction of weight loss after 16 weeks intervention by assessing early changes in hunger/satiety | Baseline, Week 4, and Week 16
  Hunger/satiety will be measured via peptide YY (PYY)
Prediction of weight loss after 16 weeks intervention by assessing early changes in hunger/satiety | Baseline, Week 4, and Week 16
  Hunger/satiety will be measured via ghrelin

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil V Dhurandhar, PhD, Principal Investigator — Texas Tech University
Locations (2):
- United States (2):
  - Texas Tech Neuroimaging Institute, Lubbock, Texas
  - Nutrition & Metabolic Health Initiative, Lubbock, Texas